CLINICAL TRIAL: NCT05753189
Title: Safety Study: A Multi-Center, Double-Masked Phase 3 Safety Study Evaluation of the Long-Term Safety of LNZ101 in Presbyopic Subjects
Brief Title: Phase 3 Safety Study for the Treatment of Presbyopia Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LENZ Therapeutics, Inc (Other)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-150-0017
Record Dates: First submitted 2023-02-07; First posted 2023-03-03 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia; Near Vision; Miosis; Eye Diseases
Keywords: Pharmaceutical Solutions; Opthalmic Solutions; Eye Drops; CLARITY; Presbyopia; Miotic
MeSH Terms: conditions — Presbyopia; Myopia; Miosis; Eye Diseases

STUDY DESIGN:
Intervention Model Description: A Multi-Center, Double-Masked Phase 3 Evaluation of the Long-Term Safety of LNZ101 in Presbyopic Subjects
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-masked treatment will be used to reduce potential of bias during data collection and the evaluation of clinical endpoints.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Combination ophthalmic solution (LNZ101) dosed bilaterally (Experimental): LNZ 101: Aceclidine/Brimonidine Ophthalmic Solution
  Interventions: Drug: Aceclidine+Brimonidine combination ophthalmic solution
- Placebo (Vehicle) ophthalmic solution dosed bilaterally (Placebo Comparator): Placebo: Proprietary Vehicle Ophthalmic Solution
  Interventions: Drug: Placebo
- Aceclidine ophthalmic solution dosed bilaterally (Experimental): LNZ 100: Aceclidine ophthalmic solution
  Interventions: Drug: Aceclidine Ophthalmic Solution

INTERVENTIONS:
Drug: Aceclidine+Brimonidine combination ophthalmic solution — Combination ophthalmic solution of Aceclidine and Brimonidine
  Other Names: LNZ101
  Arms: Combination ophthalmic solution (LNZ101) dosed bilaterally
Drug: Placebo — Placebo: Proprietary Vehicle Solution
  Other Names: Vehicle
  Arms: Placebo (Vehicle) ophthalmic solution dosed bilaterally
Drug: Aceclidine Ophthalmic Solution — Aceclidine
  Other Names: LNZ100
  Arms: Aceclidine ophthalmic solution dosed bilaterally

SUMMARY:
Safety Study of the Long-Term Safety of LNZ101 in Presbyopic Subjects

DETAILED DESCRIPTION:
Safety Study: Multi-Center, Double-Masked Phase 3 Evaluation of the Long-Term Safety of LNZ101 in Presbyopic Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent and sign a Health Information Portability and Accountability Act (HIPAA) form prior to any study procedure being performed;
2. Be able and willing to follow all instructions and attend all study visits;
3. Be 45-75 years of age of either sex and any race or ethnicity at Visit 1;
4. Be presbyopic in both eyes as determined by manifest refraction documented at Visit 1;
5. Have +1.00 to -4.00 diopter(D) of sphere calculated in minus cylinder (up to 2.00D of cylinder) in both eyes determined by manifest refraction documented at Visit 1

Exclusion Criteria:

1. Be a female of childbearing potential who is currently pregnant, nursing, or planning a pregnancy;
2. Have known contraindications or sensitivity to the use of any of the study medications or their components;
3. Have an active ocular infection at Visit 1 (bacterial, viral, or fungal), positive history of an ocular herpetic infection, preauricular lymphadenopathy, or ongoing, active ocular inflammation in either eye;
4. Have moderate or severe dry eye defined as total corneal fluorescein staining at Visit 1;
5. Have clinically significant abnormal lens findings during dilated slit-lamp biomicroscopy and fundus exam at Visit 1

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 7 visits over a total duration of approximately 28 weeks
  Percentage of subjects who experience adverse events and monocular BCDVA changes at 4m.

CONTACTS AND LOCATIONS:
Overall Officials: Alisyn Facemire, BA, Study Director — LENZ Therapeutics
Locations (36):
- United States (36):
  - Site #326, Dothan, Alabama
  - Site #302, Chandler, Arizona
  - Site #320, Mesa, Arizona
  - Site #321, Phoenix, Arizona
  - Site #328, Phoenix, Arizona
  - Site #338, Scottsdale, Arizona
  - Site #331, Sun City, Arizona
  - Site #303, Garden Grove, California
  - Site #313, Glendale, California
  - Site #334, La Jolla, California
  - Site #322, Newport Beach, California
  - Site #306, Petaluma, California
  - Site #337, Rancho Cordova, California
  - Site #304, Santa Barbara, California
  - Site #308, Littleton, Colorado
  - Site #316, Danbury, Connecticut
  - Site #319, Crystal River, Florida
  - Site #309, Mt. Dora, Florida
  - Site #317, Rock Island, Illinois
  - Site #301, Overland Park, Kansas
  - Site #307, Pittsburg, Kansas
  - Site #324, Louisville, Kentucky
  - Site #336, Alexandria, Minnesota
  - Site #330, Kansas City, Missouri
  - Site #335, Bozeman, Montana
  - Site #310, Fargo, North Dakota
  - Site #332, West Fargo, North Dakota
  - Site #329, Cincinnati, Ohio
  - Site #323, Powell, Ohio
  - Site #333, Eugene, Oregon
  - Site #312, Cranberry Township, Pennsylvania
  - Site #315, Memphis, Tennessee
  - Site #311, Smyrna, Tennessee
  - Site #314, El Paso, Texas
  - Site #327, San Antonio, Texas
  - Site #318, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No